CLINICAL TRIAL: NCT00543894
Title: Antibiotic Therapy for Hospital-Acquired Infections in ICU Patients. A Prospective, Observational, Multicenter Study (ANTHICUS)
Brief Title: Antibiotic Therapy for Hospital-Acquired Infections in ICU Patients
Acronym: ANTHICUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: SRP-HB-MER-2005/1
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2007-06

CONDITIONS: Infection in ICU
Keywords: Antibiotic, ICU, hospital acquired infection.
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Antibiotic Therapy for Hospital-Acquired Infections in ICU Patients. A prospective, observational, multicenter study (ANTHICUS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hospital-acquired infections and hospitalised in the ICU at one moment of their hospital stay
* Hospital-acquired infections accounting for eligibility are:

  * nosocomial pneumonia (including ventilator-associated pneumonia)
  * bacteremia
  * intra-abdominal infections
  * urosepsis

Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-02

SECONDARY OUTCOMES:
the frequency of appropriate antibiotic therapy (defined as the use of antibiotic(s) with "in vitro" efficacy against the identified pathogens responsible for the infection)
the frequency of "the strategy of de-escalation" according to the culture results

CONTACTS AND LOCATIONS:
Overall Officials: Pr Vogelaers, Principal Investigator — UZ Gents